CLINICAL TRIAL: NCT06953947
Title: A Comparison Between Interscalene and Costoclavicular Blocks for Pain Relief After Shoulder Surgery
Brief Title: Interscalene Versus Costoclavicular Blocks for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Muhammed Halit Tekeci, MD, Anesthesiology and Reanimation Specialist, M.D., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-16214662-050.01.04-176689116
Record Dates: First submitted 2025-04-05; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain; Shoulder Surgeries Operations; Regional Anesthesia; Costoclavicular Block; Interscalene Blocks
Keywords: analgesia; brachial plexus; postoperative pain; shoulder surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: A total of 62 patients undergoing for shoulder surgery under general anesthesia between 01.11.2022 and 01.11.2023 were divided into two groups following written informed consent, with one group receiving ISB and the other group receiving CCB. A blinded researcher recorded pain scores at postoperative 0.5, 1, 6, 12, 18, and 24 hours
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinded researcher recorded pain scores at postoperative 0.5, 1, 6, 12, 18, and 24 hours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group CCB (Experimental): The group of patients which received costoclavicular block
  Interventions: Procedure: Costoclavicular block; Drug: Costoclavicular block
- Group ISB (Experimental): The group of patients which received interscalene block
  Interventions: Procedure: Interscalene block; Drug: Interscalene Nerve Block

INTERVENTIONS:
Procedure: Costoclavicular block — The costoclavicular block was first described by Karmakar et al. in 2015. It is a type of brachial plexus block that targets the three cords located lateral to the axillary artery within the costoclavicular space. The costoclavicular space is defined as the area between the middle third of the clavicle and the anterior thoracic wall. Within this space, the cords of the brachial plexus are situated lateral to the axillary artery, positioned between the pectoralis major, subclavius, and serratus anterior muscles.
  In contrast to the traditional infraclavicular approach, the cords in the costoclavicular block are located more superficially and are more consistently clustered lateral to the axillary artery, which may facilitate visualization and needle targeting. After the needle is placed between the three cords under ultrasound guidance, the local anesthetic (20 mL of 0.25% bupivacaine) is injected.
  Arms: Group CCB
Procedure: Interscalene block — Originally described by Etienne in 1925, the technique was later refined into its modern clinical form by Alon Winnie in 1970. The interscalene approach, primarily preferred for shoulder surgeries, aims to target the upper roots of the brachial plexus (C5-C7). In interscalene block, a needle is placed under ultrasound guidance around the upper and middle trunks of the brachial plexus, which pass through the space between the anterior and middle scalene muscles, and the local anesthetic (20 mL of 0.25% bupivacaine) is injected while its spread is observed.
  Arms: Group ISB
Drug: Costoclavicular block — In costoclavicular block, the course of the three cords of the brachial plexus is visualized under ultrasound guidance, adjacent to the brachial artery beneath the clavicle. Subsequently, after the needle is placed under ultrasound guidance between the three cords, 20 mL of 0.25% bupivacaine is injected as the local anesthetic.
  Arms: Group CCB
Drug: Interscalene Nerve Block — In interscalene block, using an ultrasound probe placed on the neck, the course of the brachial plexus trunks between the anterior and middle scalene muscles is visualized. Then, after the needle is inserted under ultrasound guidance between the anterior and middle scalene muscles, 20 mL of 0.25% bupivacaine is injected as the local anesthetic.
  Arms: Group ISB

SUMMARY:
AIM: Shoulder surgeries are among the most painful surgical procedures in orthopedic practice. Interscalene brachial plexus block, although the most commonly utilized regional anesthesia technique for alleviating pain following shoulder surgery, may result in complications such as hemidiaphragmatic paresis, hoarseness. More distal blocks along the brachial plexus may provide postoperative analgesia while potentially having less effect on respiratory functions. The aim of this study is to determine whether there are differences in postoperative pain scores and opioid consumption between interscalene block (ISB) and costoclavicular brachial plexus block (CCB).

MATERIALS AND METHODS: Following ethical approval, all eligible patients undergoing for shoulder surgery under general anesthesia between 01.11.2022 and 01.11.2023 will be enrolled and to be divided into two groups following written informed consent, with one group receiving ISB and the other group receiving CCB. A blinded researcher will record pain scores at postoperative 0.5, 1, 6, 12, 18, and 24 hours. Demographic data of patients, postoperative opioid consumption, time to first analgesic request, rescue analgesic requirements, adverse effects and hemodynamic parameters will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral shoulder surgery
* ASA (American Society of Anesthesiology) class I, II and III patients

Exclusion Criteria:

* Coagulopathy
* Chronic Pulmoner Disease
* Hypersensitivity to local anesthetics
* Ipsilateral neurological deficits
* Non-communicative patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Measurement | Measured at Postoperative 0.5, 1, 6, 12, 18, and 24 hours
  The pain measurements of the patients after surgery which evaluated with visual analogue scale (VAS), ranging from 0 to 10 while 0 describes no pain at all and 10 describes the most severe pain a person can experience.

SECONDARY OUTCOMES:
Postoperative Opioid Consumption | Postoperative 24 hours.
  The total amount of opioid analgesics used which measured by the patient controlled analgesia (PCA) device for the postoperative 24 hours
Time to first analgesic request | Postoperative 24 hours
  The period of time which describes the patient's first postoperative analgesic request.
Rescue analgesic requirements | Postoperative 24 hours
  The drugs that used for additinoal analgesia.
Adverse effects | Postoperative 24 hours
  Any adverse effects related to anesthetic and analgesic procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided